CLINICAL TRIAL: NCT04851587
Title: Empowering the Management of Pain-Obesity-Weight Through Enhanced Reward
Brief Title: EMPOWER: Empowering the Management of Pain-Obesity-Weight Through Enhanced Reward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202002133-N; 1R21AG070642-01 (NIH)
Record Dates: First submitted 2021-04-01; First posted 2021-04-20 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: Back Pain; Obesity; Aging; Overweight
MeSH Terms: conditions — Low Back Pain; Back Pain; Obesity; Overweight | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-Person (or Remote) Intervention Visits (Experimental): Participants will initially complete a baseline assessment assessing study eligibility. The intervention includes 8 core in-person group sessions and 8 optional in-person group sessions (1.5 hours each) targeting standard weight loss and pain treatment content and eight individual phone calls (30 minutes each) focusing primarily on increasing environmental reward and positive affect. Intervention sessions may be delivered online through protected health information (PHI) Zoom. Group sessions will be delivered every-other week and phone calls will occur every-other week (during weeks with no group). Sessions will be administered by a study interventionist with bachelors- or masters-level training and certification in health education or a related field (e.g., Certified Health Education Specialist), and materials will be developed to be appropriate for delivery by this level of training, given the potential for greater availability of these types of health professionals.
  Interventions: Behavioral: In-Person (or Remote) Intervention

INTERVENTIONS:
Behavioral: In-Person (or Remote) Intervention — Participants will be asked to engage in self-administered activities during the intervention including pleasant activity scheduling, values clarification, mindfulness practice, goal setting, standard pain coping skills, and weight management including nutrition education and physical activity monitoring.

SUMMARY:
The central objective of research is to examine the feasibility and acceptability of an 8-month single-arm behavioral intervention (i.e., EMPOWER) among overweight/obese middle-aged and older adults with moderate-to-high impact low back pain. Intervention content will focus on standard behavioral weight loss treatment and cognitive-behavioral pain coping therapy with a focus on environmental reward and positive affect.

DETAILED DESCRIPTION:
Chronic low back pain (cLBP) is the leading cause of disability worldwide and is one of the top reasons for seeking healthcare. High-impact low back pain is particularly problematic, defined as chronic pain accompanied by significant restrictions in work, social, and/or self-care activities for six months or more. High-impact pain is associated with greater pain-related disability, opioid use, and healthcare costs compared to pain of lower impact. Thus, efforts to reduce chronic pain impact have become a public health initiative. Low back pain and overweight/obesity are highly comorbid; overweight and obese individuals are up to 43% more likely to have cLBP compared to normal weight individuals. Together, the additive effects of overweight/obesity and chronic pain may play a larger role in increasing the risk for other adverse health-related comorbidities.

The aim of this exploratory study is to examine the feasibility and acceptability of an integrated pain and weight management intervention (EMPOWER) for middle-aged and older adults with moderate-to-high impact low back pain by addressing mechanisms of environmental reward and positive affect. Forty adults (ages 45-80 years) with comorbid overweight/obesity (BMI≥25 kg/m2) and moderate-to-high impact cLBP will be assigned to an 8-month intervention, whereby they will receive a group- and telephone-based program featuring integrated behavioral weight loss treatment and cognitive-behavioral pain coping therapy. To address the key mechanisms of environmental reward and positive affect, the proposed intervention will incorporate systematic pleasant activity scheduling and values-clarification techniques. Assessments will be conducted at baseline and at the 4- and 8-month time points.

ELIGIBILITY:
Inclusion Criteria:

* 45-80 years of age
* Have a BMI≥25kg/m2
* Endorse pain in the lower back region (i.e., space between the lower posterior margin of the rib cage and the horizontal gluteal fold), knees, or hips
* Pain must occur on at least 50% of the days in the previous six months
* Pain must be rated, at minimum, of moderate intensity (rating of 3 on a numeric rating scale ranging from 0-10)
* Pain impact must be rated as moderate to severe
* Study physician reviews medical record and declares patient medically appropriate for exercise protocol

Exclusion Criteria:

* Current participation in another psychological treatment or structured weight loss program
* Severe psychiatric illness not adequately controlled by medication or other conditions anticipated to impair intervention engagement (e.g., substance abuse/dependence)
* Presence of chronic, malignant pain (e.g., cancer)
* Significant cognitive impairment (<26) on the Montreal Cognitive Assessment (MoCA)
* Inability to read and write English
* Currently undergoing radiation or chemotherapy for cancer
* Self-reported cardiac event in the past 6 months or self-reported Heart Failure (CHF)
* Currently pregnant or breastfeeding, or planning to become pregnant during the study time period
* Back, knee, or hip surgery within the past six months of study entry (or planned surgical interventions for pain during forecasted study participation)
* If currently taking prescription analgesic or psychotropic medication, must be stabilized on these treatments for >4 weeks prior to the baseline assessment
* Blood pressure higher than 180/100 mm Hg at baseline assessment
* Has had bariatric surgery in the past year or is planning to have it in the next year
* If participant reports the presence of systemic inflammatory disease (e.g., rheumatoid arthritis), the study physician will be consulted to determine eligibility

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Bartley, Ph.D, Principal Investigator — University of Florida; Megan A McVay, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McVay MA, Scotti K, Cheong J, McGargill S, Anton SA, Bartley EJ. Addressing co-occurring chronic pain and obesity simultaneously in a behavioral intervention: a pilot trial. Pilot Feasibility Stud. 2026 Jan 31. doi: 10.1186/s40814-026-01764-3. Online ahead of print. PMID 41620768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this single-arm clinical trial began in November 2021, with the last participant enrolled in January 2023. Participants with chronic musculoskeletal pain were recruited via the University of Florida Health System's clinical and administrative database. Additionally, patients were approached after their appointments at a a specialty spine clinic, and referrals were made from spine clinic providers. Recruitment took place at UF Health in the Gainesville and Jacksonville area.
Pre-assignment Details: Of the 132 individuals who expressed interest in the study and completed prescreening, 37 participants were eligible and enrolled. Of the 37 individuals who were enrolled, 33 participants commenced treatment.
Groups:
- Empower Intervention: Participants will initially complete a baseline assessment assessing study eligibility. The intervention includes 8 core in-person group sessions and 8 optional in-person group sessions (1.5 hours each) targeting standard weight loss and pain treatment content and eight individual phone calls (30 minutes each) focusing primarily on increasing environmental reward and positive affect. Intervention sessions may be delivered online through protected health information (PHI) Zoom. Group sessions were delivered every-other week and phone calls will occur every-other week (during weeks with no group).
  Participants were asked to engage in self-administered activities during the intervention including pleasant activity scheduling, values clarification, mindfulness practice, goal setting, standard pain coping skills, and weight management including nutrition education and physical activity monitoring.
Period: Overall Study
Arm/Group | Empower Intervention
Started | 37
Received the Intervention | 33
Completed | 19
Not Completed | 18
Not completed — Lost to Follow-up | 18

BASELINE CHARACTERISTICS:
Population: Consented and started the intervention
Arm/Group | Empower Intervention
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 19
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Session-level Engagement (NOTE: This is a Pilot Study and There is Not a True Primary Outcome. There Are Several Descriptive Outcomes That Will Inform Our Decision to Proceed to a Traditional, Fully Powered Clinical Trial).
Description: Treatment Engagement Questionnaire: 6-item study-adapted questionnaire assessing perceptions of engagement, interest in the session content, and usefulness of the home activities. Items are rated on a 0 to 8 scale with the mean value across sessions calculated. The total scale is create by taking the mean of the items, and has a possible range of 0 (minimum) to 8 (maximum) score. There are no subscales. Higher scores indicate greater treatment engagement.
Time Frame: Assessed at each session (every other week) up to 8 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empower Intervention
Number analyzed (Participants) | 19
score on a scale | 6.9 (1.2)

2. Primary Outcome: Global Treatment Engagement
Description: Number of participants who completed the intervention (defined as attending the final group session)
Time Frame: Baseline to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Empower Intervention
Number analyzed (Participants) | 33
Participants | 25

3. Primary Outcome: Participant Satisfaction
Description: A single treatment satisfaction item ("In an overall, general sense, how satisfied are you with the intervention program you received?"). This item was rated on a 1 to 4 scale, with a higher score indicating greater satisfaction with the treatment.
Time Frame: Month 4
Population: all assessed at 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Person (or Remote) Intervention Visits
Number analyzed (Participants) | 26
units on a scale | 3.5 (0.66)

4. Primary Outcome: Participant Satisfaction
Description: as for outcome 3
Time Frame: Month 8
Population: Those completing 8 month assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empower Intervention
Number analyzed (Participants) | 19
score on a scale | 3.7 (0.45)

5. Primary Outcome: Treatment Credibility
Description: Treatment Expectation Questionnaire: 7-item study-developed questionnaire assessing the credibility and reasonableness of the intervention. Items are rated on a 0 to 10 scale. A mean score was calculated for the questionnaire. Higher scores were indicative of greater treatment credibility.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Empower Intervention
Number analyzed (Participants) | 33
score on a scale | 7.8 (1.3)

6. Primary Outcome: Enrollment Rate
Description: Percentage of participants who enroll that commence treatment.
Time Frame: Baseline to Week 1
Population: Those who were eligible and consented
Measure: Count of Participants; unit: Participants
Arm/Group | Empower Intervention
Number analyzed (Participants) | 37
Participants | 33

7. Primary Outcome: Enrollment Rate
Description: Number of participants enrolled per week during active recruitment.
Time Frame: 63 Weeks
Measure: Mean (Standard Deviation); unit: participants enrolled per week
Arm/Group | Empower Intervention
Number analyzed (Participants) | 33
participants enrolled per week | 0.52 (0.90)

8. Primary Outcome: Participant Retention
Description: Percentage of enrolled participants who complete the 8-month time-point.
Time Frame: Baseline to 8 Months
Population: All who commence treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Empower Intervention
Number analyzed (Participants) | 33
Participants | 19

9. Secondary Outcome: Body Weight Change
Description: Kilograms weight change from baseline to 4 months measured by digital scale
Time Frame: 4 months
Population: Completed 4 month assessment
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Empower Intervention
Number analyzed (Participants) | 26
kilograms | -2.89 [-4.61 to -1.16]

10. Secondary Outcome: Pain Impact Change
Description: Research Task Force Impact Stratification Questionnaire: 9-items derived from the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form assessing pain intensity, pain interference with normal activities, and functional status. Impact stratification scores range from 8 (mild impact) to 50 (severe impact), with higher scores indicative of greater pain impact.Score represents change from baseline to 4 month assessment.
Time Frame: 4 months
Population: Those completing 4 month assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Empower Intervention
Number analyzed (Participants) | 26
score on a scale | -4.0 [-6.77 to -1.31]

11. Secondary Outcome: Pleasant Activity Engagement
Description: Percentage of pleasant activity goals met based on standardized self-report at the beginning of each phone session. Participants were queried on whether they achieved their weekly goal with the following response options (yes, no, partially). Frequencies for goal attainment were conducted, with percentage of goals met calculated across participants.
Time Frame: Baseline to 8 Months
Population: Percentage of participants meeting partial or full weekly pleasant activity engagement goals.
Measure: Number; unit: percentage of participants
Arm/Group | In-Person (or Remote) Intervention Visits
Number analyzed (Participants) | 26
percentage of participants
  Full Goals Met | 64.7
  Partial Goals Met | 28.0

12. Secondary Outcome: Meaningful Activity Participation Change
Description: Meaningful Activity Participation Assessment Questionnaire: 28-item checklist reflecting common activities that are meaningful to older adults. Items are rated both for how much time is spent on activities and how meaningful the activities are perceived to be. Items are rated on a 1 to 7 scale for frequency of activities and on a 1 to 5 scale for meaningfulness (summative values calculated). Meaningful Activity Participation Assessment scores can range from 0 to 672. Higher scores indicate greater frequency and meaningfulness of activities. Change from baseline to 4 months
Time Frame: 4 months
Population: Those completing 4 month survey
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Empower Intervention
Number analyzed (Participants) | 26
score on a scale | 6.36 [-28.20 to 40.92]

13. Secondary Outcome: Global Treatment Engagement
Description: Number of participants who completed the intervention (defined as attending the final 8 month treatment session)
Time Frame: Baseline to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Empower Intervention
Number analyzed (Participants) | 33
Participants | 17

ADVERSE EVENTS:
Time Frame: 8 months
Description: Description of adverse event conforms to clinical trials .gov definition. Data was collected non-systematically.
Arm/Group | In-Person (or Remote) Intervention Visits
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04851587/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04851587/ICF_002.pdf